CLINICAL TRIAL: NCT03474874
Title: Human Repeated Insult Patch Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeXtGen Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NNAU01-001
Record Dates: First submitted 2018-03-15; First posted 2018-03-23 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-05

CONDITIONS: Dermatitis; Allergy; Contact Allergy
MeSH Terms: conditions — Dermatitis; Hypersensitivity; Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Collagen Dressing and Comparator (Other): NeoMatriX Collagen Dressing and Comparators - positive control and normal saline will be applied to the absorbent pad portion of the exclusive dressing.
  Interventions: Device: NeoMatriX Collagen Dressing

INTERVENTIONS:
Device: NeoMatriX Collagen Dressing — Collagen wound dressing

SUMMARY:
Repeated insult patch test on healthy males and females to determine potential contact irritation or contact allergy in the skin

ELIGIBILITY:
Inclusion Criteria:

* Adults;
* Subjects must understand and execute an Informed Consent Form that includes a HIPAA statement;
* Subjects must be considered dependable and able to follow directions

Exclusion Criteria:

* Subjects who are in ill health;
* Subjects who are taking medications other than birth control;
* Female subjects who are pregnant (return positive urine pregnancy test), planning to become pregnant or lactating during the course of the trial;
* Subjects who have a history of adverse reactions to personal care products, or known sensitivity to the test materials or their constituents including patch materials;
* Subjects with any active skin disease;
* Subjects who have heavy alcohol consumption;
* Subjects with current use or history of repeated use of street drugs;
* Subjects with a significant past medical history to potentially effect results of study;
* Subjects with immunization less than 10 days prior to the test patch application;

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Consumer Product Testing Company, Inc., Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collagen Dressing and Comparator
Started | 68
Completed | 54
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Collagen Dressing and Comparator
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 59
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 46 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Erythema at the Patch Test Site is Evaluated for Each Participant
Description: Erythema Scoring Scale with 0 being no visible erythema and 5 being bullous reaction.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: erythema score
Groups:
- NeoMatriX: NeoMatriX Collagen Dressing: Collagen wound dressing
- Positive Control: 0.4% SLS on absorbent pad of occlusive dressing
- Negative Control: Normal saline on absorbent pad of occlusive dressing
Arm/Group | NeoMatriX | Positive Control | Negative Control
Number analyzed (Participants) | 54 | 54 | 54
erythema score | 0.00 [0 to 0] | 0.59 [0 to 1] | 0.00 [0 to 0.5]

2. Secondary Outcome: Sensitization Reactions
Description: Erythema Scoring Scale with 0 being no visible erythema and 5 being bullous reaction.
  Allergic Dermal Sensitization Potential - Erythema will be evaluated at the patch site for only the test material (positive and negative control will not be evaluated). Sensitization reactions will be determined at the patch test site after a two week rest period for each participant (similar to a "wash-out period"). The patch test site will be tested on the same study subject population, but using a virgin test site.
Time Frame: 5 weeks
Population: Only the experimental material (NeoMatriX) was tested for potential sensitization reactions.
Measure: Mean (Full Range); unit: erythema score
Arm/Group | NeoMatriX | Positive Control | Negative Control
Number analyzed (Participants) | 54 | 0 | 0
erythema score | 0 [0 to 0] |  |

ADVERSE EVENTS:
Time Frame: 40 days
Arm/Group | Collagen Dressing and Comparator
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT03474874/Prot_SAP_001.pdf